CLINICAL TRIAL: NCT01803178
Title: The Effect of Plant Sterols on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FDS-SCC-0574
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-02

CONDITIONS: Vascular Diseases; Hypercholesterolemia
Keywords: vascular function; plant sterols; blood lipids
MeSH Terms: conditions — Vascular Diseases; Hypercholesterolemia | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant Sterols (Active Comparator): Plant Sterols
  Interventions: Dietary Supplement: Plant Sterols
- Placebo Product (Placebo Comparator): Placebo Product
  Interventions: Dietary Supplement: Placebo Product

INTERVENTIONS:
Dietary Supplement: Plant Sterols
  Arms: Plant Sterols
Dietary Supplement: Placebo Product
  Arms: Placebo Product

SUMMARY:
The main aim of the study is to investigate, in humans, the effect of plant sterols on vascular function by measuring flow-mediated dilation (FMD).

This study also aims to study the effect of plant sterols on pulse wave velocity (PWV), aortic augmentation index (Aix), central blood pressure (CBP), office blood pressure (BP), blood lipids and plasma plant sterol concentration. At last, the effects of plant sterols on z-scores of circulating biomarkers of endothelial dysfunction and low-grade inflammation will be assessed.

For all study outcomes, effect sizes and 95% confidence intervals will be estimated.

Hypothesis: Based on available evidence, it is hypothesized that plant sterols modestly increase FMD.

DETAILED DESCRIPTION:
Plant sterols are well known for their LDL-cholesterol lowering benefit. Elevated cholesterol and especially LDL-cholesterol concentrations are established risk factors for coronary heart disease (CHD) and reducing these concentrations by dietary modification or drug treatment have been shown to reduce the risk of CHD. Direct evidence supporting a reduced risk of CHD has so far not been generated. Investigating the effects of consuming plant sterols on intermediate risk factors beyond cholesterol-lowering is therefore warranted.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and post-menopausal women
* BMI ≥ 18 and ≤ 30 kg/m2.
* Aged between 40 - 65 years.
* Having elevated LDL-cholesterol concentrations at screening (130-190 mg/dL or 3.4-4.9 mmol/L).
* Blood pressure, heart rate, haematological and clinical chemical parameters within the normal reference range as judged by the research physician

Exclusion Criteria:

* Having (previous) cardiovascular event(s) (stroke, TIA, angina, myocardial infarction, heart failure), systemic inflammatory conditions or diabetes mellitus.
* Use of over-the-counter and prescribed medication which may interfere with study measurements (i.e. statins, ezetimibe, fibrates, diabetic drugs, ARB and ACE inhibitors), to be judged by the Principal Investigator.
* Use of medical treatment for elevated TG concentrations.
* Use of antibiotics in the three months prior to screening.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months prior to screening and/or during the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation | At baseline (after 4 weeks run-in period) and after 12 weeks intervention

SECONDARY OUTCOMES:
Change in pulse wave velocity | At baseline (after 4 weeks run-in period) and after 12 weeks intervention

OTHER OUTCOMES:
Change in blood lipids | At baseline (after 4 weeks run-in period) and after 4, 8 and 12 weeks intervention
Change in plasma plant sterols | At baseline (after 4 weeks run-in period) and after 4, 8 and 12 weeks intervention
Change in plasma biomarkers of endothelial dysfunction and low-grade inflammation | At baseline (after 4 weeks run-in period) and after 12 weeks intervention
Change in aortic augmentation index | At baseline (after 4 weeks run-in period) and after 12 weeks intervention
Change in central blood pressure | At baseline (after 4 weeks run-in period) and after 12 weeks intervention
Change in office blood pressure | At baseline (after 4 weeks run-in period) and after 12 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wieneke Koppenol, MSc, Study Director — Unilever Research & Development
Locations (1):
- Charité Research Organisation, Berlin, Germany

REFERENCES:
- [Derived] Ras RT, Fuchs D, Koppenol WP, Schalkwijk CG, Otten-Hofman A, Garczarek U, Greyling A, Wagner F, Trautwein EA. Effect of a plant sterol-enriched spread on biomarkers of endothelial dysfunction and low-grade inflammation in hypercholesterolaemic subjects. J Nutr Sci. 2016 Dec 6;5:e44. doi: 10.1017/jns.2016.40. eCollection 2016. PMID 28620471
- [Derived] Ras RT, Koppenol WP, Garczarek U, Otten-Hofman A, Fuchs D, Wagner F, Trautwein EA. Increases in plasma plant sterols stabilize within four weeks of plant sterol intake and are independent of cholesterol metabolism. Nutr Metab Cardiovasc Dis. 2016 Apr;26(4):302-9. doi: 10.1016/j.numecd.2015.11.007. Epub 2015 Dec 12. PMID 26806045
- [Derived] Ras RT, Fuchs D, Koppenol WP, Garczarek U, Greyling A, Keicher C, Verhoeven C, Bouzamondo H, Wagner F, Trautwein EA. The effect of a low-fat spread with added plant sterols on vascular function markers: results of the Investigating Vascular Function Effects of Plant Sterols (INVEST) study. Am J Clin Nutr. 2015 Apr;101(4):733-41. doi: 10.3945/ajcn.114.102053. PMID 25809853